CLINICAL TRIAL: NCT05714358
Title: The Effect Of Mobile Traınıng Applıcatıons On Chronıc Renal Faılure Progressıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, ARZU KAVALA, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mobile Traınıng Applıcatıons
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Kidney Diseases, Chronic
Keywords: Chronic renal failure; mobile application; patient education
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study, the experimental and control groups were determined as 110 individuals, 55 each.
Who Masked: Participant
Masking Description: * Being chronic renal failure (stage 3)
  * Being between the ages of 18-65
  * Knowing how to read and write
  * Being able to use a smart phone
  * Volunteering to participate in the study
  * Not having a mental problem
  * Not having a communication problem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Experimental): Face to face education programme and mobile app were used.
  Interventions: Behavioral: Education
- CONTROL GROUPS (No Intervention): Only face to face education was used.

INTERVENTIONS:
Behavioral: Education — * The patients were given face-to-face training on nutrition, physical activity and drug use in chronic renal failure .
  * After the training, the biochemical parameters of the patients were followed for 6 months.
  * In this process, the questions asked by the patients in order not to hinder their right to receive information were answered.
  Arms: INTERVENTION GROUP

SUMMARY:
The purpose of research that Mobile Education Application is to evaluate its effects on the progress of chronic renal failure . The sample of the study, which is conducted with a semi-experimental design, consisted of 100 patients (50 interventions and 50 controls) who applied to the nephrology outpatient clinic of a City Hospital affiliated to the Istanbul Provincial Health Directorate. Patient Diagnosis Form, Diet Information of Hemodialysis Patients, Dietary Behavior of Hemodialysis Patients, Cognitive Behavioral Physical Activity scale and mobile education application were used as data collection tools. In the analyses of data; descriptive analyses, parametric and non-parametric tests, generalized linear mixed model and linear regression analysis are used. Firstly, face-to-face training was given to the experimental and control groups. Subsequently, a mobile education application was installed on the phones of the experimental group. The patients in the experimental group were followed for six months with the mobile education application. The content of the mobile education application; education, nutritional contents, measurement values and ask me a question sections. With the reminder system in the application, notifications were sent to the patients 2 days a week. The characteristics of the participants in both groups of the study were similar.

DETAILED DESCRIPTION:
This research; The limitations of mobile education applications to the progression of chronic renal failure were performed as a semi-treatment in order to ensure that the patients' management of their own disease was effective.Research; It was held between 01.06.2021 and 30.03.2022 in a City Hospital affiliated to Istanbul Provincial Health Directorate.The population of the study consisted of chronic renal failure stage 3 patients. Power analysis was performed using the G*Power (v3.1.9) program to determine the size of the study. The power of the study is expressed as 1-β (β = probability of type II error) and in general studies should have 80% power. When a large (d=0.8) effect size was predicted in the comparisons between groups, it was calculated that at least 26 groups were required to obtain 80% power at α=0.05 diameter. However, considering that there may be cells that can be separated from the research of maintaining its reliability and continuing the study, the experimental and control groups were determined as 110 individuals, 55 each.

İnclusion Criteria for Research

* Being chronic renal failure stage (stage 3)
* Being between the ages of 18-65
* Knowing how to read and write
* Being able to use a smart phone
* Volunteering to participate in the study
* Not having a mental problem
* Not having a communication problem

Exclusion Criteria

* Being chronic renal failure stage 1-2-4-5
* Being illiterate
* Not using a smartphone

Dependent variables: Biochemical parameters, amounts of consumed food ingredients, dietary information, behavioral and cognitive behavioral physical activity scale scores, physical activity type and duration, measurement values, eGFR value Arguments: Mobile education app

İNTERVENTİONS GROUPS FIRST INTERVIEW

* Written informed consent was obtained from patients before data were collected.
* Data; Patient identification form was collected with Diet Information of Hemodialysis Patients, Dietary Behavior of Hemodialysis Patients, Cognitive Behavioral Physical Activity scale
* The results of the biochemical parameters requested by the physician were recorded.
* The patients were given face-to-face training on nutrition, physical activity and drug use in chronic renal failure
* After the training, the mobile training application, including the training, was installed on the patient's phone, and how to use it was explained.
* Our kidneys and their functions, chronic kidney failure and its stages, nutrition in chronic kidney failure, physical activity and drug use trainings, heart rate, physical activity, blood sugar, blood pressure measurement follow-ups, content values of foods and amount of fluid consumed in the mobile education application. There was a question section and reminder systems.
* The education of the patients was followed by the researcher through the mobile education application interface.
* The patients' biochemical parameters and use of mobile education applications were followed for 6 months.
* Reminders about their education, nutritional status, physical activities and drug use were made at regular intervals (2 times a week).
* Patients were able to reach the researcher whenever they wanted from the ask me a question section of the mobile application.

SECOND INTERVIEW

* The results of the biochemical parameters requested by the physician were recorded.
* Data collection forms were filled out again by interviewing the patients over the phone.

CONTROL GROUPS FIRST INTERVIEW

* Written informed consent was obtained from patients before data were collected.
* Data; Patient identification form was collected with Diet Information of Hemodialysis Patients, Dietary Behavior of Hemodialysis Patients, Cognitive Behavioral Physical Activity scale
* The results of the biochemical parameters requested by the physician were recorded.
* The patients were given face-to-face training on nutrition, physical activity and drug use in chronic renal failure .
* After the training, the biochemical parameters of the patients were followed for 6 months.
* In this process, the questions asked by the patients in order not to hinder their right to receive information were answered.

SECOND INTERVIEW

* The results of the biochemical parameters requested by the physician were recorded.
* Data collection forms were filled out again by interviewing the patients over the phone.

ELIGIBILITY:
Inclusion Criteria:

Being chronic renal failure (stage 3)

* Being between the ages of 18-65
* Knowing how to read and write
* Being able to use a smart phone
* Volunteering to participate in the study
* Not having a mental problem
* Not having a communication problem

Exclusion Criteria:

Being chronic renal failure stage 1-2-4-5

* Being illiterate
* Not using a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Patient Information Form: | Basaline
  This form developed by the researcher; sociodemographic characteristics of the patient (age, gender, educational status), disease and treatment data (primary diagnosis, disease stage, other disease states), height, weight, Body Mass Index (BMI), daily amount of fluid consumed, amount of urine, medication using status and laboratory findings (urea, uric acid, creatinine, sodium, potassium, calcium, phosphorus, parathormone, albumin, iron, glucose, total cholesterol, HDL, LDL, triglyceride, urine amount, hemoglobin, hematocrit, eGFR and blood pressure value). ) consists of.

SECONDARY OUTCOMES:
Dietary Knowledge Scale of Hemodialysis Patients (HHDB): | Baseline
  It was developed by Bulantekin Düzalan and Çınar in 2014. The Cronbach's alpha reliability coefficient of the scale is 0.86 and 0.73, respectively. The scale is a 3-point Likert scale. For the knowledge scale, the participants were asked to answer each item as "True, False, I don't know". In the knowledge scale, correct is scored as "1", incorrectly as "0" and I do not know "0". The lowest is 0 and the highest is 18 points. The cut-off point of the scale was 7, and it was evaluated as "good knowledge level" over 7 points. There is no reverse scored item in the scale.
Dietary Knowledge Scale of Hemodialysis Patients (HHDB): | 6 months later
  It was developed by Bulantekin Düzalan and Çınar in 2014. The Cronbach's alpha reliability coefficient of the scale is 0.86 and 0.73, respectively. The scale is a 3-point Likert scale. For the knowledge scale, the participants were asked to answer each item as "True, False, I don't know". In the knowledge scale, correct is scored as "1", incorrectly as "0" and I do not know "0". The lowest is 0 and the highest is 18 points. The cut-off point of the scale was 7, and it was evaluated as "good knowledge level" over 7 points. There is no reverse scored item in the scale.

OTHER OUTCOMES:
Dietary Behavior Scale of Hemodialysis Patients (HHDD): | Baseline
  It was developed by Bulantekin Düzalan and Çınar in 2014. The Cronbach's alpha reliability coefficient of the scale is 0.86 and 0.73, respectively. The scale is a 5-point Likert type scale. For the Attitude and Behavior Scale, the participants were asked to answer each item as "I strongly disagree, I disagree, I am undecided, I agree, I totally agree". In the behavior scale, it is scored as "1" to strongly disagree, "2" to disagree, "3" to undecided, "4" to agree and "5" to completely agree. The lowest score is 13 and the highest 65 points. The cut-off point of the scale was 46, and it was evaluated as "good behavior" over 46 points. There is no reverse scored item in the scale.
Dietary Behavior Scale of Hemodialysis Patients (HHDD): | 6 months later
  It was developed by Bulantekin Düzalan and Çınar in 2014. The Cronbach's alpha reliability coefficient of the scale is 0.86 and 0.73, respectively. The scale is a 5-point Likert type scale. For the Attitude and Behavior Scale, the participants were asked to answer each item as "I strongly disagree, I disagree, I am undecided, I agree, I totally agree". In the behavior scale, it is scored as "1" to strongly disagree, "2" to disagree, "3" to undecided, "4" to agree and "5" to completely agree. The lowest score is 13 and the highest 65 points. The cut-off point of the scale was 46, and it was evaluated as "good behavior" over 46 points. There is no reverse scored item in the scale.
Cognitive Behavioral Physical Activity Scale (BDFA): | Baseline
  The scale was developed by Schembre et al. in 2015 and its Turkish validity and reliability was performed by Eskiler et al. in 2016. The scale consists of 3 sub-dimensions and 15 questions. It is a 5-point Likert type scale with the form of '1' Strongly Disagree and '5' Strongly Agree. It includes three sub-factors as outcome expectation, self-regulation, and personal barriers. Outcome expectation = (1 + 2+ 9 + 13 + 14) / 5, self-regulation = (3 + 4 + 5 + 6 + 8) / 5, personal barriers = (7 + 10 + 11 + 12 + 15) / 5 , total score = Expectation of Outcome + Self-Regulation - Personal Barriers. A high score indicates a good level. The maximum score that can be obtained from the scale is nine.
Cognitive Behavioral Physical Activity Scale (BDFA): | 6 months later
  The scale was developed by Schembre et al. in 2015 and its Turkish validity and reliability was performed by Eskiler et al. in 2016. The scale consists of 3 sub-dimensions and 15 questions. It is a 5-point Likert type scale with the form of '1' Strongly Disagree and '5' Strongly Agree. It includes three sub-factors as outcome expectation, self-regulation, and personal barriers. Outcome expectation = (1 + 2+ 9 + 13 + 14) / 5, self-regulation = (3 + 4 + 5 + 6 + 8) / 5, personal barriers = (7 + 10 + 11 + 12 + 15) / 5 , total score = Expectation of Outcome + Self-Regulation - Personal Barriers. A high score indicates a good level. The maximum score that can be obtained from the scale is nine.
Mobile Education Application (Application) | for 6 months
  The application name was determined as 'Live with Your Own Kidney'. With the mobile application, the amount of food and liquid consumed by the patients, blood pressure measurements, pulse, blood sugar measurements, physical activity and drug use were followed for 6 months. With the Ask me a question section, patients were able to reach the researcher 24/7 and ask questions. With the application, reminders were given to the patients in the form of short messages 2 days a week. The effect of the mobile application on the course of the disease was evaluated by monitoring the nutrition and measurement values of the patients with apply.

CONTACTS AND LOCATIONS:
Locations (1):
- Arzu Kavala, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No